CLINICAL TRIAL: NCT03865927
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial of GKT137831 in Patients with Idiopathic Pulmonary Fibrosis
Brief Title: GKT137831 in IPF Patients with Idiopathic Pulmonary Fibrosis
Acronym: GKT137831
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Temple University (Other); Tulane University (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Steven R. Duncan, MD, PI, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-300001635
Record Dates: First submitted 2019-03-01; First posted 2019-03-07 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Reactive oxygen species (ROS); nicotinamide adenine dinucleotide phosphate (NADPH) oxidase
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — setanaxib

STUDY DESIGN:
Intervention Model Description: Following screening assessments, IPF patients who meet all inclusion/exclusion criteria will be randomly assigned to receive one of the following treatments in a ratio of 1:1:
  • Arm A (n=30) - GKT137831 Treatment:
  GKT137831 will be administered orally, at a dose of 400 mg bid, for a total of 24 weeks.
  • Arm B (n=30) - Placebo Treatment:
  Arm B subjects will receive matching placebo for the same duration.
  Participants will be followed in face-to-face visits with trial personnel every 6 weeks for 24 weeks to assess drug effects and monitor safety during their treatments, and by phone surveillances one month thereafter.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GKT137831 (Experimental): GKT137831 will be administered orally, at a dose of 400 mg twice daily, for a total of 24 weeks.
  Interventions: Drug: GKT137831
- Placebo Oral Tablet (Placebo Comparator): Identically-appearing placebo oral tablets will be administered orally, twice daily, for a total of 24 weeks.
  Interventions: Other: Placebo Oral Tablet

INTERVENTIONS:
Other: Placebo Oral Tablet — see Arm/Group description
  Arms: Placebo Oral Tablet
Drug: GKT137831 — GKT137831 is a NOX enzyme inhibitor
  Arms: GKT137831

SUMMARY:
A placebo-controlled, multicenter, randomized trial to test GKT137831 in ambulatory patients with idiopathic pulmonary fibrosis. This drug is an inhibitor of nicotinamide adenine dinucleotide phosphate (NADPH) oxidase (NOX) isoforms. The investigators hypothesize the drug will decrease pulmonary injury due to reactive oxygen species (ROS) generated by NOX enzymes, which are believed to play an important role in the development of IPF. Treatment with GKT137831 could result in significant benefit for a lung disease that has, until now, been almost invariably inexorable.

This clinical trial represents the bedside application of a series of NOX translational and basic studies and discoveries, over several years, from the laboratory of Dr. Victor Thannickal.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40-85 years old.
2. A diagnosis of IPF that fulfills current American Thoracic Society (ATS) Consensus Criteria.
3. IPF duration <5 years, based on the date of definitive diagnosis.
4. Ability and willingness to give informed consent and adhere to study requirements.
5. Ratio of forced expiratory volume in 1 second to forced vital capacity (FEV1/FVC) >70% of predicted values

Exclusion Criteria:

1. Diagnosis of major comorbidities expected to interfere with study participation
2. History of malignancy, excluding basal or squamous cell skin cancer and low-risk prostate cancer, the latter defined as stage T1 or T2a, with prostate specific antigen <10 ng/dl. NOX inhibition is not known to promote cancer, and these criteria are within current guidelines.
3. The occurrence of any acute infection requiring systemic antibiotic therapy within 2 weeks prior to Screening (Visit 1).
4. Treatment for >14 days within the preceding month with >20 mg. prednisone (or equivalent) or any treatment during the last month with a cellular immunosuppressant (e.g., cyclophosphamide, methotrexate, calcineurin inhibitors, etc.), given increased risks of opportunistic infections.
5. Treatment with any investigational agent within 4 weeks of Screening (Visit 1) or 5 half-lives of the investigational medicinal product (whichever is longer).
6. Fertile women who do not agree to contraception or abstinence, or who are breast feeding. IPF is a disease of older adults, and male predominant, so this will not be a frequent consideration.
7. Subjects with known hypersensitivity to GKT137831 or its excipients (e.g. capsule "bulking" agents).
8. A history of bone marrow disorder including aplastic anemia, or marked anemia defined as hemoglobin < 10.0 g/dL (or 6.2 mmol/L).
9. Severe cardiovascular disease, defined as any of the following within the preceding 12 weeks: acute myocardial infarction or unstable angina, a coronary revascularization procedure, congestive heart failure (NYHA Class III or IV), or stroke, including a transient ischemic attack.
10. Evidence of cardiac conducting abnormalities, defined as second or third degree atrial-ventricular (AV) block not successfully treated with a pacemaker, or a personal or family history of long QT syndrome (QTc interval >450 msec for males or 470 msec for females).
11. End-stage renal disease requiring dialysis.
12. Undergoing transplantation evaluation, or listed with the United Network for Organ Sharing (UNOS) as a lung transplantation candidate at the time of enrollment in this trial.
13. Liver function tests (transaminases, alkaline phosphatase, direct and total bilirubin) >3x upper limit of normal values

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Surrogate biomarker of oxidative stress by mass spectroscopy | From baseline thru week 24
  Changes in concentrations of circulating o,o'-dityrosine, as determined by mass spectroscopy in plasma, in terms of absolute concentrations and percentages of baseline, will be compared within and between treatment arm participants.

SECONDARY OUTCOMES:
Collagen degradation product by enzyme linked immunoabsorbant assay | Baseline to week 24
  Changes in concentrations of the collagen degradation product, serum C1M measured by enzyme linked immunsorbent assays will be compared between baseline values and those at 24 weeks, and between experimental arm and control participants.
Pulmonary function by spirometry | Baseline to week 24
  Forced vital capacity (FVC), measured by spirometer at baseline, will be compared to values at the conclusion of the study and between the two treatment arms.
Ambulatory ability by measuring walk distance in six minutes | Baseline to week 24
  Six-minute walk distance (6MWD) will be compared at baseline and as changes from baseline among experimental arm participants and control subjects
Evaluation of safety by adverse events | Baseline to week 24
  The number and severity of adverse events will be compared between experimental arm participants and those in the control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Duncan, MD, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Tulane University Medical Center, New Orleans, Louisiana
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Temple University Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No